CLINICAL TRIAL: NCT04684680
Title: Effect of Zamzam Water on Amniotic Fluid Index, in Oligohydramnios : a Randomized Controlled Trial
Brief Title: The Role of Zamzam Water in Idiopathic Oligohydramnios
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aswu/3oo/6/19
Record Dates: First submitted 2020-09-05; First posted 2020-12-24 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Oligohydramnios
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Intervention Model Description: open label randomized controlled trial
Masking Description: open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zamzam water (Experimental): patient will receive the normal need of daily requirement of water (2.5 liter) in form of zamzam water till patients deliver or till term
  Interventions: Dietary Supplement: zamzam water
- tap water (Active Comparator): will receive the normal need of daily requirement of water (2.5 liter) in form of tap water
  Interventions: Dietary Supplement: tap water

INTERVENTIONS:
Dietary Supplement: zamzam water — will receive the normal need of daily requirement of water (2.5 liter) in form of zamzam water till patients deliver or till term
  Other Names: study group
  Arms: zamzam water
Dietary Supplement: tap water — will receive the normal need of daily requirement of water (2.5 liter) in form of tap water
  Other Names: Active Comparator
  Arms: tap water

SUMMARY:
The aim of this study is to evaluate the efficacy of drinking zamzam water versus tap water in increasing the AF index in women with oligohydramnios.

DETAILED DESCRIPTION:
Oligohydramnios refers to decrease in amniotic fluid and it is defined as a deepest fluid pocket of less than 2 cm or an amniotic fluid index of 5 cm or less. Oligohydramnios complicates 0.5% to 8% of pregnancies, and 12 % if postdates When it occurs in first half of pregnancy it is associated with birth defects while in second half it causes poor fetal growth, malpresentations , FHR decelerations , MAS , Fetal suicidal syndrome and increases cesarean section and management and prognosis depend on gestational age

ELIGIBILITY:
Inclusion Criteria:

* pregnant female with idiopathic oligohydramnios

Exclusion Criteria:

* patients with medical disorder
* congenital anomalies
* premature rupture of membrane
* Patient refuse to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant female with idiopathic oligohydramnios
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
amniotic fluid index | 10 weeks
  the change of the amniotic fluid volume

CONTACTS AND LOCATIONS:
Overall Officials: nahla w shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No